CLINICAL TRIAL: NCT02514252
Title: A Preliminary Study of Sublingual Fentanyl for the Management of Breakthrough Pain Analgesia in Patients With Advanced Cancer
Brief Title: Sublingual Fentanyl for the Management of Breakthrough Pain
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: INSYS Therapeutics Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-0264; NCI-2015-01447 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2015-07-31; First posted 2015-08-03 (Estimated); Results first posted 2021-05-18 (Actual); Last update posted 2021-05-18 (Actual); Status verified 2021-04

CONDITIONS: Advanced Cancers
Keywords: Advanced Cancers; Metastatic; Recurrent cancer; Incurable cancer; Fentanyl sublingual spray; FSS; Questionnaires; Surveys; Mental ability tests; Phone calls; Study diary; Pain control
MeSH Terms: conditions — Neoplasm Metastasis; Recurrence; Agnosia | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Fentanyl Sublingual Spray (FSS) (Experimental): Hospitalized participants asked to complete a number of surveys at baseline. Participants then receive one single dose of intravenous opioid rescue for their first episode of breakthrough pain, and then receive up to 4 doses of FSS for subsequent episodes of breakthrough pain. Initial FSS starting dose is proportional to the patient's morphine equivalent daily dose (MEDD). Symptom questionnaire completed at baseline and after last dose of FSS while hospitalized. Mental ability tests given while hospitalized 30 minutes after first dose of current pain medication, and 30 minutes after each FSS dose. At the time of discharge, if FSS was helpful in controlling participant's pain, they are then able to continue with FSS use for 1 month. Participants given study diary to document pain level, how many times FSS used, and any side effects experienced each day.
  Interventions: Drug: Fentanyl Sublingual Spray (FSS); Behavioral: Questionnaires; Behavioral: Mental Ability Tests; Behavioral: Study Diary

INTERVENTIONS:
Drug: Fentanyl Sublingual Spray (FSS) — Stage 1: First Pain Episode - Single dose of breakthrough opioid given from existing PCA pump equivalent to 10% of their MEDD.
  Second Pain Episode - Single dose of FSS equivalent to 16-32% of MEDD. If not effective at 30 minutes, participant repeats same dose one more time (with a cap of 1600 mcg total; i.e. dose given 30 minutes ago + dose now = 1600 mcg maximum.
  Third Pain Episode (at least 4 hours after second episode) - Participant required 2 breakthrough FSS doses for the last episode of breakthrough pain, or if the effective dose has not been identified, he/she will double the last administered dose. If breakthrough pain not effective at 30 minutes, participant repeats same dose one more time (with a cap of 1600 mcg total; i.e. dose given 30 minutes ago + dose now = 1600 mcg maximum).
  Stage 2: If FSS successful in hospital, upon discharge, FSS used as first choice of pain medication instead of oral pain medication for pain for up to 4 weeks.
  Other Names: Fentanyl SL Spray
Behavioral: Questionnaires — Symptom questionnaire completed at baseline and after last dose of FSS while hospitalized. After Day 28, questionnaire completed over the phone about participant's opinion of research study.
  Other Names: Surveys
Behavioral: Mental Ability Tests — Mental ability tests given while hospitalized 30 minutes after first dose of current pain medication, and 30 minutes after each FSS dose.
Behavioral: Study Diary — Participants given study diary to document pain level, how many times FSS used, and any side effects experienced each day.

SUMMARY:
The goal of this clinical research study is to learn if an investigational dose of fentanyl sublingual spray (FSS) can help to control pain in patients with advanced cancer when given in an outpatient and inpatient setting.

DETAILED DESCRIPTION:
Study Visits and Study Drug Administration:

This study has 2 stages. Stage 1 will be completed while you are in the inpatient unit of the hospital and Stage 2 will be completed after you are discharged from the hospital.

Stage 1:

While you are in the hospital, if you have a pain episode, the research nurse will give you a single dose of your current pain medication from your existing infusion pump. You will then be asked to rate your current level of pain . You will also be asked if you are having any side effects at 15 minutes and at 30 minutes after the dose has been administered. You will also complete the 4 tests of mental abilities after about 30 minutes.

If after 1-4 hours you have another episode of pain, you will be given a single dose of FSS. You will spray FSS under your tongue and hold it there for about 30-60 seconds before swallowing. You will be asked about your current level of pain at about 15 minutes and 30 minutes after your dose of FSS. You will also complete the 4 tests of mental abilities after about 30 minutes. If you do not feel any pain relief after 30 minutes, you will spray FSS 1 more time under your tongue and you will repeat the pain and mental ability tests.

If you still do not feel any pain relief after about 4 hours from the last dose of FSS, you will spray a double dose of FSS under your tongue up to 2 times and your pain level and mental abilities will be tested at 15 and 30 minutes after each dose.

You may receive FSS up to 4 times total while you are in the hospital.

After your last dose of FSS, you will complete a questionnaire about how your symptoms are after receiving FSS. This should take about 2 minutes to complete.

End of Stage 1:

If FSS was able to help you control your pain, you will stop taking FSS and go back to receiving your regular pain medication for the rest of your hospital stay. When you are discharged from the hospital, you will continue on to Stage 2 of the study (described below) to receive FSS for up to 4 weeks at home. Before you are sent home, you will also be prescribed pain medication to take in addition to the FSS, if needed. Your doctor will explain how to take this medication before you are discharged.

If FSS was not able to help control your pain, your participation in this study will end and you will continue to be treated with standard pain medications.

Stage 2:

If you are taking part in Stage 2, you will use FSS as your first choice of pain medication instead of oral pain medication for pain for up to 4 weeks. At any time that you have a pain episode, you will spray FSS under your tongue.

You will always have the choice of using the pain medication your doctor prescribed to you as a backup every 2 hours as needed for pain. However, it is very important that you do NOT use the oral pain medications at the same time as FSS. If you still have pain after taking FSS, you must wait at least 2 hours before using your pain medications. After 2 more hours if you have another episode of pain, you may use another dose of FSS for pain relief.

Do not take more than 4 doses of FSS each day.

You will be given a patient diary to write down each day your pain level, how many times you used FSS, and any side effects you may have. You will be called at least 2 times each week by a member of the study staff to discuss your diary and to answer any questions you may have. The study staff will also ask you which pain medication you are using besides FSS, how easy you think it is to use FSS, how effective you think FSS is, and how satisfied you are with your current pain medications. Each phone call should last about 10 minutes.

After Day 28, you will complete a questionnaire over the phone about your opinion of this research study. This should take about 5 minutes to complete.

Length of Study:

Your active participation in this study is over after you complete the last questionnaire. You will be taken off study if intolerable side effects occur or if you are unable to follow study directions.

Follow-Up:

About 30 days after your study visit, you will be called by the study staff and asked how you are feeling and about any side effects you may be having. This call should last about 10 minutes.

This is an investigational study. FSS is FDA approved and commercially available for the treatment of pain in cancer patients. It is considered investigational to use the dose of FSS used in this study and to use FSS both in inpatient and outpatient settings.

About 30 participants will be enrolled in this study. All will take part at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with advanced cancer (locally advanced, metastatic, recurrent and/or incurable cancer).
2. Opioid tolerant, taking daily doses of strong opioid pain medication in the past 1 week.
3. On strong opioid intravenous continuous infusion MEDD >=70 mg/day at the time of enrollment.
4. Inpatient at MD Anderson seen by palliative care team.
5. Background cancer pain that is <=3/10 in the last 24 hours.
6. Breakthrough cancer pain that is >=4/10 in the last 24 hours.
7. Stable pain control defined as rescue doses <=6 in last 24 hours.
8. Age >=18
9. Ability to communicate in English

Exclusion Criteria:

1. Memorial Delirium Assessment Scale >13/30
2. History of opioid abuse
3. CAGE positivity (>=2/4)
4. Allergy to fentanyl
5. Grade 2 or higher oral mucositis
6. Unable/unwilling to sign consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2016-02-02 (Actual); Primary Completion 2019-11-04 (Actual); Study Completion 2019-11-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suresh Reddy, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with advanced cancers aged >=18 years were recruited from MD Anderson Center.
Groups:
- Fentanyl Sublingual Spray (FSS): Fentanyl sublingual spray was administered with a starting dose of 100 mcg up to 1600 mcg maximum for each breakthrough pain.
Period: Overall Study
Arm/Group | Fentanyl Sublingual Spray (FSS)
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Fentanyl Sublingual Spray (FSS)
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 6
Marital status [Count of Participants; unit: Participants]
  Married | 5
  Separated/Divorced | 1
Education [Count of Participants; unit: Participants]
  Some high School | 1
  Some College | 2
  Completed College | 2
  Did not answer | 1
Cancer Type [Count of Participants; unit: Participants]
  Colon | 2
  Gastric | 1
  Melanoma | 1
  Cholangiocarcinoma | 1
  Lymphoma | 1

OUTCOME MEASURES:

1. Primary Outcome: Effective Dose of Fentanyl Sublingual Spray (FSS)
Description: To determine the effective dose of Fentanyl sublingual spray in the management of breakthrough pain (4 episodes) in hospitalized patients with advanced cancer receiving continuous opioid infusion in which the first starting dose would be proportional to the patients Morphine Equivalent Daily Dose. It will use Alberta Breakthrough Pain assessment tool with 15 questions.
Time Frame: Up to 1 months after discharge from the hospital
Population: Data was not collected due to low accrual and early termination.
Arm/Group | Fentanyl Sublingual Spray (FSS)
Number analyzed (Participants) | 0

2. Secondary Outcome: Difference Between Intravenous Opioid and Fentanyl Sublingual Spray
Description: To estimate the differences in the pain response between intravenous opioid breakthrough and fentanyl sublingual spray at effective dose. Pain will be assessed in a 0-10 numeric rating scale that assesses pain intensity now, where 0=no pain at all, and 10=worst possible.
Time Frame: Up to 1 month after discharge from the hospital
Population: Data was not collected due to low accrual and early termination.
Arm/Group | Fentanyl Sublingual Spray (FSS)
Number analyzed (Participants) | 0

3. Secondary Outcome: Safety, Tolerability, Pattern of Use and Efficacy
Description: To determine the safety, tolerability, pattern of use and efficacy of Fentanyl sublingual spray in patients with advanced cancer
Time Frame: Up to 1 month after discharge from the hospital
Population: Data was not collected due to low accrual and early termination.
Arm/Group | Fentanyl Sublingual Spray (FSS)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 24 hours after taking fentanyl sublingual spray
Arm/Group | Fentanyl Sublingual Spray (FSS)
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 3/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fentanyl Sublingual Spray (FSS) (N=6)
Drowsiness (Nervous system disorders) | 3
Nausea (Gastrointestinal disorders) | 1
Itching (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-12-16): https://cdn.clinicaltrials.gov/large-docs/52/NCT02514252/Prot_SAP_000.pdf